CLINICAL TRIAL: NCT04275453
Title: Comparison of the Short-Term Effect of Dietary Carbohydrate Restriction Versus Exogenous Ketone Supplementation on Myocardial Glucose Suppression and Timing to Achieve a State of Ketosis Using FDG PET/CT Serial Imaging
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 834253
Record Dates: First submitted 2020-01-06; First posted 2020-02-19 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketogenic diet - 24 hours (Experimental): Subjects will undergo FDG PET/CT after 1 day of dietary modification (ketogenic diet for at least 3 meals) and 12 hours of fasting prior to FDG injection.
  Interventions: Drug: FDG; Other: Ketogenetic Diet
- Ketogenic diet - 72 hours (Experimental): Subjects will then undergo FDG PET/CT after 3 day of dietary modification (ketogenic diet for at least 9 meals) and 12 hours of fasting prior to FDG injection.
  Interventions: Drug: FDG; Other: Ketogenetic Diet
- Exogenous ketone ester (Experimental): Subjects will undergo FDG PET/CT after 1 dose of ketone drink administration after 12 hours of fasting prior to FDG injection. The dosing of ketone drink administration (approximately 65 mL) will be weight based (714 mg/kg), which is crucial to replicating ketone levels between participants. The KE drink will be administered approximately 45 minutes prior to FDG injection as concentrations of ~3 mmol/L are reached within 60 minutes . By way of comparison, website marketing of the commercial drink recommends ingestion 30 minutes prior to athletic performance. We will also perform echocardiography immediately before and 30 minutes after the drink.
  Interventions: Drug: FDG; Dietary Supplement: Ketone Drink

INTERVENTIONS:
Drug: FDG — FDG is a FDA approved radiotracer which each subject will have 3 positron emission tomography/computed tomography (PET/CT) scan performed.
Dietary Supplement: Ketone Drink — Subjects will undergo FDG PET/CT after 1 dose of ketone drink administration after 12 hours of fasting prior to FDG injection. The dosing of ketone drink administration (approximately 65 mL) will be weight based (714 mg/kg), which is crucial to replicating ketone levels between participants
  Arms: Exogenous ketone ester
Other: Ketogenetic Diet — Subjects needs to be on Ketogenetic diet
  Arms: Ketogenic diet - 24 hours; Ketogenic diet - 72 hours

SUMMARY:
The purpose of this study is to test different methods of preparation that can be used prior to a test called an FDG PET/CT scan. FDG PET/CT scans are routinely done for evaluation of heart inflammation. Standard preparation for the scan includes a ketogenic (high fat and low carbohydrate) diet for 24 hours and overnight fasting to help suppress the amount of sugar taken up in the heart muscle. However, Investigator still do not know if this preparation is the most effective method. So the Investigator, want to investigate alternative methods for decreasing the amount of sugar uptake seen in the heart during FDG PET/CT scan, thus, investigator will have participants try up to 3 different methods of preparation prior to the FDG PET/CT scans to see which type of preparation works the best.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, at least 18 years of age
2. No history of cardiovascular disease, including hypertension, hyperlipidemia, coronary artery disease, cardiac surgery, arrhythmias per medical record review and/or self-report
3. No history of diabetes mellitus, chronic liver or kidney disease per medical record review and/or self-report.
4. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine or serum pregnancy test before the first study visit.
2. Inability to tolerate imaging procedures in the opinion of the investigator or treating physician.
3. Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-01-05 (Estimated); Study Completion 2023-01-05 (Estimated)

PRIMARY OUTCOMES:
Comparing the myocardial glucose suppression in Ketogenetic diet vs. external Ketone supplement by looking at the FDG uptake using PET/CT | 3 years
  Comparing the myocardial glucose suppression in Ketogenetic diet vs. external Ketone supplement by looking at the FDG uptake using PET/CT. Images will be qualitative and semi-quantitatively assessed. The entire right and left ventricular walls will be contoured in a dedicated nuclear medicine workstation (MIM Software) to create volume of interest s(VOI) and derive the maximum and mean standardized uptake value (SUV) and total glycolytic activity (TGA), all measures of glucose utilization. Blood pool activity within the left ventricular cavity will be used as reference. Complete myocardial suppression will be defined as FDG activity (by any measure) in the left ventricular wall lower than blood pool activity in the ventricular cavity.

SECONDARY OUTCOMES:
The optimal duration of ketosis to produce myocardial suppression by looking at the FDG uptake using PET/CT by comparing the data out of 1 day keto diet Arm versus 3 days Keto diet Arm | 3 years
  The optimal duration of ketosis to produce myocardial suppression by looking at the FDG uptake using PET/CT by comparing the data out of 1 day keto diet Arm versus 3 days Keto diet Arm.
Understanding the relationship between serum β-hydroxybutyrate (BHB) levels and myocardial glucose by looking at the FDG uptake using PET/CT by comparing the data out of keto diet Arm versus Ketone supplement Arm. | 3 years
  Understanding the relationship between serum β-hydroxybutyrate (BHB) levels and myocardial glucose by looking at the FDG uptake using PET/CT by comparing the data out of keto diet Arm versus Ketone supplement Arm by measuring serum levels of BHB, free fatty acid, acylcarnitine, glucose, and insulin at each FDG PET/CT visit. Approximately 15 mLs of blood will be drawn and used to measure B-Hydroxybutyrate (BHB), acylcarnitines, insulin, glucose and free fatty acid and other targeted metabolomics
comparing the transthoracic echocardiogram changes before and after the Ketone supplement drink to assess the effect of Ketone supplement | 3 years
  comparing the transthoracic echocardiogram changes before and after the Ketone supplement drink to assess the effect of Ketone supplement. Transthoracic Echocardiogram: Ultrasound will be used to create an image of the internal parts of the heart. This test is being done to assess any changes in cardiac function with the ketone drink. We will perform echocardiography before and approximately 30 minutes after the drink.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No